CLINICAL TRIAL: NCT02796638
Title: Adaptive Servo-Ventilation In Acute Heart Failure Patients Protecting the Heart
Brief Title: Adaptive Servo-Ventilation In Acute Heart Failure Patients Protecting the Heart and Kidneys
Acronym: ASLEEP PK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: ResMed Foundation (Other)
Responsible Party: Principal Investigator, Nancy Gardetto, Ph.D, Research Scientist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H150082
Record Dates: First submitted 2016-06-06; First posted 2016-06-13 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Sleep Apnea, Obstructive
Keywords: Acute Heart Failure; Positive-Pressure Ventilation; Adaptive Servo-Ventilation
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minute Ventilation Adaptive Servo-Ventilation plus SOC (Experimental): Patients in this arm will be instructed to use the adaptive servo-ventilation (ASV) device for up to five days of inpatient stay while in the hospital. Patients are encouraged to use the device during any and all hours of sleep, and as needed during waking hours. Apart from this treatment, no other interventions will be administered, and the patient's standard of care will not otherwise be altered for the purposes of the study.Two 6-mL tubes of blood will be drawn once daily for up to 5 days, and daily questionnaires will be administered regarding sleep and health quality.
  Interventions: Device: Adaptive Servo-Ventilation
- Standard of Care (SOC) (No Intervention): Patients in this arm will not have their standard of care as dictated by their provider altered in any way. Two 6-mL tubes of blood will be drawn once daily for up to 5 days, and daily questionnaires will be administered regarding sleep and health quality.

INTERVENTIONS:
Device: Adaptive Servo-Ventilation — A positive pressure airway device that increases and decreases inspiration pressure in concordance with the patient's natural breathing cycles.
  Arms: Minute Ventilation Adaptive Servo-Ventilation plus SOC

SUMMARY:
The primary hypothesis of this study is: the use of minute ventilation-adaptive servo-ventilation (MV-ASV) during hospitalization will mitigate deterioration in renal function and prevent kidney injury in patients admitted with acute heart failure (AHF) compared to those receiving usual care. We will validate and extend our pilot study by taking a deeper dive into the effects of ASV on diuretic dose, urine output and new and exciting biomarkers of renal function and kidney injury. If our hypothesis proves correct, it strongly suggests that ASV lessens injury to the kidney and could lead to a new paradigm for the treatment of AHF. When use of high dose of diuretics are anticipated or in whom chronic kidney disease (CKD) or acute kidney injury (AKI) is present on arrival to the Emergency Department, use of MV-ASV might decrease the amount of diuretics needed, allow for continued use of ACE inhibitors, and ultimately mitigate rises in creatinine and decreases in effective glomerular filtration. Since kidney injury is a major factor in those patients with early 30-day readmission following discharge, this therapy could become quite popular.

DETAILED DESCRIPTION:
OBJECTIVE(S): The main goal of this study is to evaluate the utility of a Minute Ventilation Adaptive Servo-ventilation (MV-ASV) device in mitigating deterioration in renal function and prevent kidney injury in patients admitted with acute heart failure compared to those receiving usual care. We will be assessing the effects of MV-ASV on diuretic dose, urine output and new and exciting biomarkers of renal function and kidney injury. If our hypothesis proves correct, it strongly suggests that ASV lessens hypoxia to the kidney and could lead to a new paradigm for the treatment of AHF. When use of high dose of diuretics are anticipated or in whom CKD or AKI is present on arrival to the Emergency Department, use of MV-ASV might decrease the amount of diuretics needed, allow for continued use of ACE inhibitors, and ultimately mitigate rises in creatinine and decreases in effective glomerular filtration. Since kidney injury is a major factor in those patients with early 30-day readmission following discharge, this therapy could become quite popular.

RESEARCH DESIGN: This is an interventional, principal investigator-initiated project with patient enrollment, cohort development and data analysis. We will recruit 66 patients with acute heart failure and evidence of volume overload and elevated BNP, since we anticipate a 10% dropout. Half will be pre-selected to have CKD with eGFR < 60 ml/min/1.73 m2. Randomization will be attempted within first six hours of hospital presentation. The participants will be randomized one of the following two groups: 1) those receiving only standard therapy or 2) those receiving standard therapy and adaptive servo-ventilation (ASV) therapy.

METHODOLOGY:

Methods:

1. Consenting of patient: every attempt will be made to consent within six hours of evaluation, as we feel there is a good window for ASV here. Maximum time to consent is 24 hours.
2. Sleep and breathing assessment: Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale, Pulmonary Sleep Lab Questionnaire, Sleep Diary, Likert Scale
3. Blood Sample Collections:
4. Two 10cc (20cc total) blood samples in standard collection tubes will be obtained via venipuncture or a peripheral IV line from each enrolled patient at the time of enrollment.
5. One sample will be collected in a lithium heparin tube and the other sample will be collected in an EDTA tube. Initial blood samples will be collected after the initiation of standard medical therapy and stabilization for acute heart failure.
6. The blood samples will be analyzed for cardiac biomarkers such as BNP, high sensitivity troponins (hsTnI), endothelin-1 (ET-1), kidney injury molecule-1 (KIM-1) by Singulex, and adrenomedullin (hADM) by Sphingotec.

   Remaining blood samples will be banked for future biomarker analysis. All samples will be held at the VASDHS in a clinical laboratory storage facility indefinitely for future analysis of biomarkers such as those of inflammation, fibrosis and cardiorenal syndrome. NO GENETIC TESTING will be done on the samples.
7. As obligated, we will report any incidental findings of FDA approved biomarkers performed, as a part of further analysis of banked specimens, to the patient through their treating physicians.
8. All specimens will be frozen at -80 degrees Celsius for storage.
9. Specimens with evidence of hemolysis will not be analyzed.
10. MV-ASV Treatment and Respiration Monitoring:

    * Adaptive Servo-Ventilation (ASV) therapy will be placed on the patient by the respiratory therapy team as soon as the patient is enrolled in the study. The ASV device will be on ASV Auto mode, which has an automatic expiratory positive airway pressure (EPAP) adjustment based on the patient's breathing. The ASV Auto default EPAP range is 4-15cmH2O with a pressure support range of 3-15cmH2O. The backup rate of the ASV is adaptive based on the patient's respiratory rate. However, if the automatic ventilation setting is not suitable to maintain target ventilation, then a setting of 15 breaths per minute will be used.
    * We will ask the patients to use the ASV therapy during all hours of sleeping during their stay in the hospital and during times when they are awake, if they feel comfortable using it.
    * The patient will be closely monitored during the first few hours to make sure the patients are comfortable, have the right settings and are without mask leaks. The monitoring team will consist of members from Cardiology, Pulmonary Critical Care and Respiratory Therapy.
11. Repeat following assessments in the hospital each day for up to five days

    * Two tubes of 10cc each (20 cc total)
    * Likert dyspnea assessment
    * Sleep diary entry once each day for up to 5 days
    * Urine outputs
    * Daily weights
    * Dose of diuretics
12. Additional hospital data to be recorded:

    * Presence of arrhythmias
    * Need for inotropes
    * Need for intubation
    * Number of ICU days
    * Total number of hospital days
    * Need for renal consult
    * Electrolytes
    * BNP
    * Troponins
13. Once the subject is discharged from the hospital, the following will happen:

    * They will be seen at 30 days for following:
    * Evaluation for events
    * Sleepiness scales: Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale, Pulmonary Sleep Lab Questionnaire, Sleep Diary, Likert Scale
    * Two tubes of blood (10cc each) will be drawn, as described above to assess renal function and AKI
    * They will not be reimbursed for this visit
14. Power analysis • The comparison of groups of size 30 and 30 has a power of 0.815 to detect an effect equal to a group difference of (0.75) standard deviations. This would apply to all variables in univariate tests at significance level of 0.05 with appropriate corrections for multiple comparisons.

CLINICAL RELATIONSHIPS: The potential benefit of this study includes the validation of the use of an ASV device in the treatment of heart failure. ASV treatment might decrease the amount of diuretics needed, allow for continued use of ACE inhibitors, and ultimately mitigate rises in creatinine and decreases in effective glomerular filtration. ASV treatment may lessen hypoxia to the kidney and could lead to a new paradigm for the treatment of AHF.

IMPACT/SIGNIFICANCE: Heart failure is a major cause of both death and healthcare spending in the United States. ASV is a cost effective, non-invasive treatment that can improve symptoms and cardiac outcomes in patients with heart failure. Validation of an MV-ASV device as an effective treatment could help improve prognosis and quality of life in patients with this often terminal condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older.
2. Admitted with a clinical diagnosis of acute heart failure.
3. Evidence of congestion (rales, JVP, CXR, edema).
4. BNP >300pg/mL
5. If BMI >35 kg/m2, then BNP >100 pg/ml.
6. Consent within 24 hours of admission, but every attempt will be made to consent within six hours.
7. Patients with known sleep disordered breathing (SDB) can be included.
8. One-half of patients in each group will have chronic kidney disease (CKD) with GFR less than 60.

Exclusion Criteria:

1. Age < 18 years.
2. Unable to provide informed consent within 24 hours of admission.
3. Current participation in a pharmaceutical or treatment-related clinical study.
4. Intubated.
5. Hypercarbic (ie. Acute Respiratory Acidosis) from reasons other than acute heart failure.
6. Cardiogenic shock.
7. Clinical diagnosis of COPD exacerbation as the primary reason for hospital admission.
8. History of non-compliance to medications and treatment.
9. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in Renal Biomarkers | 30 days post-discharge
  Mean paired change in measured blood urea nitrogen (BUN), serum creatinine (> 0.3 mg/dL increase in 48 hours), neutrophil gelatinase-associated lipocalin (NGAL), Pro-encephalin (Penkid), and endothelin

SECONDARY OUTCOMES:
Change in Renal Biomarkers | up to 90 days post-discharge
  Mean paired change in measured blood urea nitrogen (BUN), serum creatinine (> 0.3 mg/dL increase in 48 hours), neutrophil gelatinase-associated lipocalin (NGAL), Pro-encephalin (Penkid), and endothelin
Reduction in Decrease of eGFR | up to 30 days post-discharge
  A hypothesized reduction in eGFR decrease of 25% in the treatment group compared to the control group
Reduction in Decrease of eGFR | up to 90 days post-discharge
  A hypothesized reduction in eGFR decrease of 25% in the treatment group compared to the control group
Disposition and post-discharge composite events | up to 30 days post-discharge
  To assess patients for composite 30 days events, reduction of subendocardial ischemia in the hospital and at 30 days, reduction of LV wall stress and volume in the hospital and at 30 days; to assess patients for endothelial function, inflammation, and propensity toward fibrosis in the hospital and at 30 days, all of which can influence renal function.
Disposition and post-discharge composite events | up to 90 days post-discharge
  To assess patients for composite 30 days events, reduction of subendocardial ischemia in the hospital and at 90 days, reduction of LV wall stress and volume in the hospital and at 90 days; to assess patients for endothelial function, inflammation, and propensity toward fibrosis in the hospital and at 30 days, all of which can influence renal function
Other markers of renal function | up to 30 days post-discharge
  To assess patients for cumulative dose of loop diuretic, urine output, blood urea nitrogen, incidence of acute kidney injury (AKI), biomarkers of AKI, eGFR at 30 days, mean paired change in urinary biomarker levels, and serum creatinine.
Other markers of renal function | up to 90 days post-discharge
  To assess patients for cumulative dose of loop diuretic, urine output, blood urea nitrogen, incidence of acute kidney injury (AKI), biomarkers of AKI, eGFR at 30 days, mean paired change in urinary biomarker levels, and serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Gardetto, Ph.D., Principal Investigator — Veterans Affairs San Diego Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified and used only within our local research group.

REFERENCES:
- [Result] Ronco C, McCullough PA, Anker SD, Anand I, Aspromonte N, Bagshaw SM, Bellomo R, Berl T, Bobek I, Cruz DN, Daliento L, Davenport A, Haapio M, Hillege H, House A, Katz NM, Maisel A, Mankad S, Zanco P, Mebazaa A, Palazzuoli A, Ronco F, Shaw A, Sheinfeld G, Soni S, Vescovo G, Zamperetti N, Ponikowski P. Cardiorenal syndromes: an executive summary from the consensus conference of the Acute Dialysis Quality Initiative (ADQI). Contrib Nephrol. 2010;165:54-67. doi: 10.1159/000313745. Epub 2010 Apr 20. PMID 20427956
- [Result] Ronco C, Cicoira M, McCullough PA. Cardiorenal syndrome type 1: pathophysiological crosstalk leading to combined heart and kidney dysfunction in the setting of acutely decompensated heart failure. J Am Coll Cardiol. 2012 Sep 18;60(12):1031-42. doi: 10.1016/j.jacc.2012.01.077. Epub 2012 Jul 25. PMID 22840531
- [Result] McCullough PA, Bouchard J, Waikar SS, Siew ED, Endre ZH, Goldstein SL, Koyner JL, Macedo E, Doi K, Di Somma S, Lewington A, Thadhani R, Chakravarthi R, Ice C, Okusa MD, Duranteau J, Doran P, Yang L, Jaber BL, Meehan S, Kellum JA, Haase M, Murray PT, Cruz D, Maisel A, Bagshaw SM, Chawla LS, Mehta RL, Shaw AD, Ronco C. Implementation of novel biomarkers in the diagnosis, prognosis, and management of acute kidney injury: executive summary from the tenth consensus conference of the Acute Dialysis Quality Initiative (ADQI). Contrib Nephrol. 2013;182:5-12. doi: 10.1159/000349962. Epub 2013 May 13. PMID 23689652
- [Result] Ng LL, Sandhu JK, Narayan H, Quinn PA, Squire IB, Davies JE, Bergmann A, Maisel A, Jones DJ. Proenkephalin and prognosis after acute myocardial infarction. J Am Coll Cardiol. 2014 Jan 28;63(3):280-9. doi: 10.1016/j.jacc.2013.09.037. Epub 2013 Oct 16. PMID 24140658